CLINICAL TRIAL: NCT03809559
Title: Repeatability and Reproducibility of Quantitative MRCP
Status: Completed | Type: Observational
Sponsor: Perspectum (Industry)
Responsible Party: Sponsor
Other Study IDs: MRCP_RR
Record Dates: First submitted 2019-01-15; First posted 2019-01-18 (Actual); Last update posted 2019-08-28 (Actual); Status verified 2018-11

CONDITIONS: Primary Sclerosing Cholangitis; Primary Biliary Cirrhosis; Gallstones; Liver Diseases
Keywords: Magnetic Resonance Cholangiopancreatography (MRCP)
MeSH Terms: conditions — Cholangitis, Sclerosing; Liver Cirrhosis, Biliary; Gallstones; Liver Diseases | interventions — Multiparametric Magnetic Resonance Imaging

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Biliary Conditions: Participants who have a history of a biliary tree related condition
  Interventions: Device: MRCP+
- Liver conditions: Participants who have a history of a non-biliary tree related liver condition
  Interventions: Device: MRCP+
- Healthy Volunteers: Participants who have do not have a diagnosed liver condition and are in general good health
  Interventions: Device: MRCP+

INTERVENTIONS:
Device: MRCP+ — Participants will undergo an initial abdominal MRI scan in a fasted state. They will then be asked to drink 400ml pineapple juice before undergoing four further abdominal MRI scans with short breaks in between each scan.
  Other Names: Quantitative Magnetic Resonance Cholangiopancreatography; LiverMultiScan; Multiparametric MRI; MRI-PDFF; MRCP

SUMMARY:
This study aims to determine the repeatability and reproducibility of Quantitative Magnetic Resonance Cholangiopancreatography (MRCP).

Imaging scientists at Perspectum Diagnostics have developed a hessian-based mathematical model to enhance conventional MRCP to a 3D geometric model of the biliary tree, 'Quantitative MRCP'. This enables advanced quantitative measurement of bile duct width, orientation, branching point and curvative metrics.

The technology has been validated against 3D printed phantoms for accuracy, and early clinical research has demonstrated the technology has potential for clinical impact, with improvement in radiologist performance versus conventional non-enhanced MRCP imaging (Vikal et al 2017).

Quantitative MRCP aims to act as a tool to not only improve assessment of the current status of the biliary tree, but also act as a mechanism to track change within the ducts. Thus, it must be established that any change between scans is due to change in the physiology of the individual and not due to a quirk or fault of the technology.

In order to achieve this a series of scans will be performed on an individual over a short period of time, for which the condition of the biliary tree within that individual can be assumed to be constant. Between each scan, subject and coil repositioning will occur.

The study will recruit a group of adult volunteers, from both diseased groups and healthy groups in order to achieve a range of physiological biliary metrics.

DETAILED DESCRIPTION:
Biliary-related conditions, such as autoimmune conditions Primary Biliary Cholangitis (PBC), and Primary Sclerosing Cholangitis (PSC), and also cancers such as cholangiocarcinoma, affect tens of thousands of individuals in the UK each year. All biliary conditions require careful tracking of the structure and integrity of the biliary tree so that intervention can be carefully planned and with that, outcomes improved.

The current non-invasive gold-standard for assessment of the biliary tree is MRI-based Magnetic Resonance Cholangiopancreatography (MRCP). This method uses no contrast and takes up to 10 minutes to obtain within a normal scan event. However, there are several limitations to its use which include, images having great variability in quality and are used mainly for qualitative analysis. Using conventional MRCP a consultant can, depending on image quality; identify key structures, inform diagnosis, and give a general assessment on the health of the biliary tree structure. However, current MRCP imaging only allows limited quantitative assessment of the ducts. More extensive, objective quantification has the potential to dramatically improve the usability of MRCP imaging.With this in mind, imaging scientists at Perspectum Diagnostics have developed a hessian-based mathematical model to enhance conventional MRCP to a 3D geometric model of the biliary tree, 'Quantitative MRCP'. This enables quantitative measurement of bile duct width, orientation, branching point and curvative metrics.

The technology has been validated against 3D printed phantoms for accuracy, and early clinical research has demonstrated the technology has potential for clinical impact, with improvement in radiologist performance versus conventional non-enhanced MRCP imaging (Vikal et al 2017). Thus, further research into the technology and its viability as an enhancement to current procedure is necessary if it is to replace conventional MRCP as the primary method of non-invasive biliary assessment.

Integral to the development of any new technology, is demonstration of the repeatability and reproducibility of the method. This is the inter-examination variability in results. Quantitative MRCP aims to act as a tool to not only improve assessment of the current status of the biliary tree, but also act as a mechanism to track change within the ducts. Thus, it must be established that any change between scans is due to change in the physiology of the individual and not due to a quirk or fault of the technology.

The above will be tested by a series of scans performed on an individual over a short period of time, for which the condition of the biliary tree within that individual can be assumed to be constant. Between each scan, subject and coil repositioning will occur. The study will recruit a group of adult volunteers, from both diseased groups and healthy groups in order to achieve a range of physiological biliary metrics.

Quantitative MRCP is an MRI based method, requiring no contrast, however consuming a drink containing manganese improves the quality of MRCP images significantly (Frisch et al., 2017), and therefore patients are routinely asked to drink pineapple juice (naturally high in manganese) before having a clinical MRCP scan. At present, multiparametric MRI to assess the health of liver tissue is performed in a fasted state (Banerjee et al., 2014), however, in order to offer a comprehensive liver scan including both MRCP and multiparametric MRI in the same scan, it is important to understand whether consuming pineapple juice will affect the multiparametric MRI measurements of cT1, PDFF and T2*.

MRI is safe and non-invasive, with no known risks to patients as long as they are appropriately screened to ensure they have no contraindications to MRI (e.g.pacemaker, metal implant that is not certified as MR-safe).

ELIGIBILITY:
Inclusion Criteria:

* Persons over the age of 18 years
* Participant is willing and able to give informed consent for participation in the study.
* EITHER: Participant has a medical history of a liver or biliary tree related condition OR: Person is a healthy volunteer.

Exclusion Criteria:

* The participant may not enter the study if they have any contraindication to magnetic resonance imaging (inc pregnancy, extensive tattoos, pacemaker, shrapnel injury, severe claustrophobia).
* The participant may not enter the study if they have an allergy to pineapple juice.
* Any other cause, including a significant disease or disorder which, in the opinion of the investigator, may either put the participant at risk because of participation in the study, or may influence the participant's ability to participate in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Participants will be identified in one of two ways.
  * Participants who have previously taken part in one of Perspectum's ethically approved studies and consented during that study to be contacted again in the event of any future study.
  * Participants who self-identify via advertisement on Perspectum's online and social media channels, or through collaboration with the investigator's charity partners.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2018-07-19 (Actual); Primary Completion 2018-09-08 (Actual); Study Completion 2019-03-08 (Actual)

PRIMARY OUTCOMES:
Assessment of Repeatability and Reproducibility of Quantitative MRCP | 6 months
  Assessment of the variability of bile duct volume, bile duct diameter, branching points and locations of regions of variation in bile duct widths and percentages, as measured by quantitative MRCP between:
  A. Repeated scans of the same participant acquired under the same conditions
  B. Repeated scans of the same participant acquired on scanners which differ by field strength and/or manufacturer

SECONDARY OUTCOMES:
Intra and Inter-operator reproducibility | 6 months
  Statistical assessment of the agreement among quantitative MRCP analyses performed by both trained operators and expert radiologists.
Comparison of conventional MRCP and quantitative MRCP | 6 months
  Statistical assessment of the agreement between quantitative MRCP analyses (performed by both trained operators and expert radiologists) and clinician ground truth (biliary tree assessment obtained by expert radiologists using conventional MRCP)

OTHER OUTCOMES:
Assessment of the impact of pineapple juice consumption upon LiverMultiScan performance | 6 months
  Statistical assessment of the agreement among cT1, PDFF and T2* measurements before and after consuming pineapple juice.

CONTACTS AND LOCATIONS:
Overall Officials: Rajarshi Banerjee, BM BCh MSc DPhil, Principal Investigator — Perspectum Diagnostics
Locations (2):
- United Kingdom (2):
  - Addenbrookes Hospital, Cambridge, Cambridgeshire
  - Oxford Centre for Clinical Magnetic Resonance Research, Oxford, Oxfordshire

IPD SHARING:
Plan to Share IPD: No